CLINICAL TRIAL: NCT05285189
Title: The Effects of Isotonic Saline as Irrigation Fluid on Serum Electrolytes and Blood Gases in Bipolar Transurethral Resection of Prostate (TUR-P) : A Prospective Observational Study
Brief Title: Effects of Isotonic Saline As Irrigation Fluid In Transurethral Resection of Prostate (TUR-P) Operations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Assoc.Prof., Istanbul University
Other Study IDs: 2018/1378
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hyperchloremic Acidosis; Transurethral Resection of Prostate; Normal Anion Gap Metabolic Acidosis; Anesthesia
Keywords: Blood gas analysis; TUR-P; Irrigation Fluid; Hyperchloremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Benign hypertrophy of the prostate (BPH) is a disease seen in 20% of men over the age of 50 and in 40% of those over the age of 70. The gold standard in the treatment of BPH is transurethral resection of the prostate using high-frequency diathermy. Today, this process is done with the bipolar technique, in which isotonic saline (isotonic sodium chloride %0.9) is used as the irrigation fluid. This irrigation fluid, which is used after long operation and deep tissue resection, can enter the systemic circulation through the opened venous sinuses.

It has been shown in clinical studies that postoperative acute hyperchloremia (serum Cl level > 110 mmol/L) develops after the use of intravenous normal saline solution in large amounts in the perioperative period.

Our aim is to detect hyperchloremia and associated metabolic acidosis without anion gap in the follow-up of these patients. Our primary hypothesis in this study is that hyperchloremic metabolic acidosis will develop due to the high amount of normal saline used in TUR-P.

.

DETAILED DESCRIPTION:
Benign hypertrophy of the prostate (BPH) is a disease seen in 20% of men over the age of 50 and in 40% of those over the age of 70. The gold standard in the treatment of BPH is transurethral resection of the prostate using high-frequency diathermy. Today, this process is done with the bipolar technique, in which normal saline (isotonic sodium chloride %0.9) is used as the irrigation fluid. In bipolar TUR-P, resection is performed using 25000 - 30000 ml normal saline for irrigation. This irrigation fluid, which is used after long operation and deep tissue resection, can enter the systemic circulation through the opened venous sinuses.

It has been shown in clinical studies that postoperative acute hyperchloremia (serum Cl level > 110 mmol/L) develops after the use of intravenous normal saline solution in large amounts in the perioperative period. McCluskey et al. found that 30-day mortality, prolonged hospital stay, and postoperative renal dysfunction developed in patients who received perioperative intravenous normal saline and subsequently developed acute hyperchloremia. Megan E. et al. Scheingraber et al. reported that the use of normal saline increases the risk of acidosis and kidney damage, also compared Ringer's lactate and normal saline infusion in patients who underwent gynecological surgery and showed that hyperchloremic metabolic acidosis developed in normal saline group. Excessive and rapid administration of normal saline solution by parenteral route causes hyperchloremic metabolic acidosis, which adversely affects the organism. According to recent studies, the development of hyperchloremic metabolic acidosis increases the cost and mortality, prolongs the hospitalization period, and causes renal dysfunction.

Our aim is to detect hyperchloremia and associated metabolic acidosis without anion gap in the follow-up of these patients. Our primary hypothesis in this study is that hyperchloremic metabolic acidosis will develop due to the high amount of normal saline used in TUR-P.

The investigators expect that an increase in the amount of fluid, prolongation of the operation time, and capsule perforation will increase hyperchloremia and deepen metabolic acidosis. If it causes hyperchloremic metabolic acidosis, the contribution of the amount of irrigation fluid or the duration of the operation can be determined, and the maximum amount of fluid that does not adversely affect the organism and the duration of the operation can be predicted.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Having had a TUR-P operation
* Using of bipolar technic
* American Society of Anesthesiology (ASA) grade I-III
* Receiving patients consent

Exclusion Criteria:

* Failure to record preoperative and postoperative blood gas data
* Patient refusal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Having benign prostate hyperplasia
Study Population: * Male gender who being prostate hyperplasia
  * Having had a TUR-P operation
  * Using of bipolar technic
  * American Society of Anesthesiology (ASA) grade I-III
  * Receiving patients consent
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Serum Chlorid level | Up to 4 hours
  Chlorid level is evaluated with blood gas analysis 3 times in total, at the beginning of the operation, at the 40th minute of the operation and 1st hour of arrival in post-anesthesia care unit.

SECONDARY OUTCOMES:
Serum anion gap level | Up to 4 hours
  It is evaluated with blood gas analysis 3 times in total, at the beginning of the operation, at the 40th minute of the operation and 1st hour of arrival in post-anesthesia care unit.
Serum lactate level | Up to 4 hours
  It is evaluated with blood gas analysis 3 times in total, at the beginning of the operation, at the 40th minute of the operation and 1st hour of arrival in post-anesthesia care unit.
Presence&absence of capsule perforation during the operation | Up to 4 hours
  Effect of capsule perforation on hyperchloremia
Amount of prostate tissue resected during the operation | Up to 4 hours
  The effect of the amount of prostate tissue resected during the operation on hyperchloremia.
Amount of used normal saline for irrigation during the operation | Up to 4 hours
  The effect of the amount of used normal saline for irrigation during the operation on hyperchloremia.
Duration of operation | Up to 4 hours
  The effect of operation time on hyperchloremia.
Incidence of postoperative acute kidney injury | Up to 48 hours
  AKI was diagnosed by an increase in serum creatinine concentration >50% from a baseline creatinine concentration measured within 48 hours prior to enrollment
Incidence of mortality rate | Up to 6 months
  Mortality of the patients was screened retrospectively at 6 months postoperatively.
Length of hospital stay | Up to 1 week
  Length of patients hospital stay was screened retrospectively at 1 week postoperatively.
Number of participants with urethral stricture | Up to 6 months
  Diagnosis will be made by urethroscopy in patients with voiding complaints.
Number of participants with urinary bladder hematoma | Up to 1 week
  Urinary system ultrasound in patients with severe hematuria

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc.Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Barker ME. 0.9% saline induced hyperchloremic acidosis. J Trauma Nurs. 2015 Mar-Apr;22(2):111-6. doi: 10.1097/JTN.0000000000000115. PMID 25768968
- [Result] Dombre V, De Seigneux S, Schiffer E. [Sodium chloride 0.9%: nephrotoxic crystalloid?]. Rev Med Suisse. 2016 Feb 3;12(504):270-2, 274. French. PMID 26999998